CLINICAL TRIAL: NCT05002439
Title: Multicenter Randomized Clinical Trial to Analyze the Efficacy of a Spanish Healthcare ministRy Based In InTervention to Reduce Frailty Status in Prefrail Older Adults (FRAILMERIT)
Brief Title: RCT to Analyze the Efficacy of a Spanish Healthcare ministRy Based In InTervention to Reduce Frailty Status in Prefrail Older Adults
Acronym: FRAILMERIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Universitario de Albacete (Other)
Responsible Party: Principal Investigator, Pedro Abizanda, Principal Investigator, Complejo Hospitalario Universitario de Albacete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRAILMERIT
Record Dates: First submitted 2021-07-23; First posted 2021-08-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Frailty; Aged; Exercise
Keywords: Frailty; Aged; Multimodal training
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomization will be made by clusters, being every cluster a different Primary Care center in order to avoid contamination. Randomization on a 1:1 relationship between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group multicomponent physical exercise program, nutritional intervention and Frailty training (Experimental): Group multicomponent physical exercise program, nutritional intervention program and Primary Care training in Frailty.
  The exercise program will be delivered by trained experts in groups of 6 participants, and will be based on the recommendations presented in the Spanish Healthcare Ministry document updated 2022. This program includes balance, flexibility, and strength and power exercises. The program will be realized twice a week, during 45 minutes time, for 12 weeks, twice, with a discontinuation period of 2 months. Nutritional recommendations will de presented by a nutritionist at the beginning of the intervention to the Primary Care physicians. Primary Care Physicians will have the opportunity of referring high risk participants to their Geriatrics Department Participants when appropriate, following Healthcare Ministry algorithm
  Interventions: Other: Multicomponent physical exercise program and a nutritional intervention
- Control group (No Intervention): Control group will receive usual care by their Primary Care Physicians. Healthy lifestyle recommendations including exercise and nutritional recommendations will be offered

INTERVENTIONS:
Other: Multicomponent physical exercise program and a nutritional intervention — The exercise program will be delivered by trained experts in groups of 6 participants, and will be based on the recommendations presented in the Spanish Healthcare Ministry document. This program includes balance, flexibility, and strength and power exercises. The program will be realized twice a week, during 45 minutes time, for 16 weeks, twice a year. Nutritional intervention will be based on the results of MNA-SF. If the results of this instrument show normal nutrition status, general nutritional recommendations will de presented by a nutritionist twice a year before the physical exercise program. If MNA-SF shows nutritional risk or malnutrition, oral nutritional supplementation will be offered. Primary Care Physicians will have the opportunity of referring high risk participants to their Geriatrics Department Participants when appropriate, following Healthcare Ministry algorithm
  Arms: Group multicomponent physical exercise program, nutritional intervention and Frailty training

SUMMARY:
Objectives: The main objective is to analyze the efficacy of an intervention based on the algorithm proposed by the Spanish Healtcare Ministry (see figure in annex 1) at Primary Care level to reduce Frailty status or Physical Function in community-dwelling older adults. Secondary objectives are: 1. To analyze if the intervention is cost-effective; 2. To analyze if the intervention reduces hospitalizations and emergency department visits, incident disability, falls, institutionalization, mortality, Primary Care visits and Drug use, and improves quality of life.

Methodology: Multicentric Randomized Clinical Trial in 273 Prefrail or Frail or with a gait speed lower that 0.8 m/s community-dwelling women and men with an age equal or greater to 70 years, attended in selected Primary Care centers of Spain (Albacete, Hellín, Barcelona, Madrid, La Carlota, and Tacoronte). Randomization will be made by clusters, being every cluster a different Primary Care center in order to avoid contamination. Randomization on a 1:1 relationship between groups. The main outcome variable will be Frailty status or Physical function change (main composite outcome) at 8-month follow-up measured with the Frailty Phenotype and the Short Physical Performance Battery (SPPB) respectively. All instrumentation will follow the guidelines of the Spanish Healthcare Ministry algorithm for frailty updated 2022. Intervention will consist on a groupal multicomponent physical exercise program, a nutritional intervention program and a training in Frailty to Primary Care centers. The intervention will be delivered by trained experts in groups of 6 participants, and will be based on the recommendations of the Spanish Healthcare Ministry document, updated in 2022.

DETAILED DESCRIPTION:
Hypothesis An intervention based on the algorithm proposed by the Spanish Healtcare Ministry (see figure in annex 1) at Primary Care level will be effective in reducing Frailty status or Physical Function (composite outcome) in community-dwelling older adults.

Main Objective

To analyze the efficacy of an intervention based on the algorithm proposed by the Spanish Healtcare Ministry (see figure in annex 1) at Primary Care level to reduce Frailty status or Physical Function (composite outcome) in community-dwelling older adults.

Secondary objectives

1. To analyze if the intervention is cost-effective 2. To analyze if the intervention reduces hospitalizations and emergency department visits 3. To analyze if the intervention reduces incident disability 4. To analyze if the intervention reduces falls 5. To analyze if the intervention reduces institutionalization 6. To analyze if the intervention improves quality of life 7. To analize if the intervention decreases mortality 8. To analyze if the intervention reduces Primary Care visits and Drug use

1. Design Multicentric Randomized Clinical Trial
2. Study subjects Prefrail or Frail or with a gait speed lower than 0.8 m/s community-dwelling women and men with an age equal or greater to 70 years, attended in selected Primary Care centers of Spain (Albacete, Hellín, Barcelona, Madrid, La Carlota, and Tacoronte).

   Sample size The sample size was calculated to find a difference between groups of 15% in the percentage of respondents (reduction in at least one frailty criteria); 25% in the intervention group (algorithm implementation) and 5% in the control group, alpha < 0.05 and power 80%. A 15% of loses will be assumed. Using the program GRANMO (https://www.imim.cat/ofertadeserveis/es_granmo.html), the number of participants per group is 82, for a total of 164 participants. However, due to COVID conditions, the sample size was increased up to 273 participants.
3. Randomization Randomization will be made by clusters, being every cluster a different Primary Care center, in order to avoid contamination. Randomization will be computer-based with a 1:1 relationship between groups. Every Primary Care center will include at least 24 participants (two Primary Care Physicians at each one). Because exercise groups will be composed of 6 participants. For these reasons, 12 Primary Care centers will be needed, 6 with intervention and 6 control
4. Instrumentation All instrumentation will follow the guidelines of the Spanish Healthcare Ministry algorithm for frailty, updated 2022.

   First, older adults attending the selected Primary Care centers (Albacete, Hellín, Barcelona, La Carlota, Tacoronte and Madrid) will receive a Barthel index assessment, a frailty phenotype assessment and a gait speed measurement in every Primary Care center. If patients present a Barthel index greater than 85 plus either a prefrailty or frailty say¡tutus or a walking speed lower than 0,8 m/s, they will be offered to entry the trial by the Primary Care Physician.

   In order to warrant the independence of recruitment, randomization of the Primary Care centers will be undertaken when a center arrives the 24 participants.

   If the center is considered "usual care", physicians will realize a baseline visit to participants, collecting all study variables, and will make healthy lifestyles recommendations.

   If the center is considered "intervention", physicians will realize a basal visit to participants collecting determined variables, and they will receive the intervention described below.

   Follow-up visits to analyze results will be conducted at 3, 5 and 8 months. Adverse events will be monitored and communicated on presentation. Monitoring will be conducted throughout the clinical trial.
5. Data collection and analysis For this project we will use the tool "Research Electronic Data Capture" (REDCap) for Electronic Data Capture (EDC), designed for creating surveys and questions using branching logic and stop actions. Some of the question will be created as a data collection instrument, and other will be selected from the data collection instruments in REDCap shared library, a repository for data collection instruments and forms. REDCap is a web-based application developed by Vanderbilt University to capture data for clinical research. REDCap uses instruments such as surveys and forms as research capture tools and is designed to provide a secure environment so that research teams can collect and store highly sensitive information. They are workflow-based and focus on collecting data and exporting it to statistical programs and other data analysis software. More information can be viewed at: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5764586/. INVESTEN, participating in the Project will provide this tool for free.

   Data will be stored for up to 15 years by the investigators. All data will be anonimyzed and stored in a secure manner. Analysis will be maid on an intention-to-treat basis by the principal investigator that will be blinded to group assignment. Risk reduction will be presented for the principal variable. Differences in secondary objectives will be analyzed with risk reductions, difference of means or proportions when convenient.
6. Economic models In order to collect information on the health and non-health resources consumption, specific questionnaires would be designed, for both, for patients as well as for caregivers. For the economic evaluation, we will perform two different analyses, a cost-effectiveness analysis (CEA) and a cost-utility analysis (CUA). The CEA will be carried out comparing both outcomes and monetary valuation of the resources used in the group of patients who receive the intervention with the control group (usual care). Thereby, the incremental cost-effectiveness ratio (ICER) reveals the cost per unit of benefit of switching from usual care to the intervention group. The health results measured by the ICER would be the following: Frailty status change, hospitalization, incident disability, and falls. Furthermore, CUA is a special type of cost-effectiveness analysis that uses the Quality-Adjusted Life-Year (QALY) as outcome.

   Both CEA and CUA would be conducted separately considering both the societal perspective (that is, all costs included) and the National Health System perspective (taking into consideration healthcare costs and costs related to the intervention).

   Additionally, several univariate sensitivity analysis as well as probabilistic sensitivity analysis will be carried out in order to test how sensitive the results obtained from the ICER and the ICUR are when varying both costs and health results.
7. Ethics The Study has been approved by the Ethics Review Committee of Albacete (February meeting), and will be presented to the rest of local Ethics Committees. The information form for participants and informed consent is presented in the annexes. There have been two amendments to the first approved version, that were approved by the ethics committee, V3 in 2023 and the final V4 in 2025.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults with age equal or greater than 70 years.
* Barthel index > 85
* Gait speed < 0.8 m/s OR frailty /prefrailty using the frailty phenotype
* Ability to realize the physical exercise program
* Capacity to understand the procedures and interventions of the trial
* Capacity to understand and sign the informed consent

Exclusion Criteria:

* Major contraindications for exercise: Severe aortic valve stenosis, myocardial infarction in the previous 6 weeks, Venous thromboembolic disease in the previous 6 weeks.
* Inability to conduct the physical tests of the trial
* Inability to understand the procedures of the trial
* Active solid organ or hematologic neoplasm other than basocellular skin neoplasm, or life expectancy lower than one year.
* Surgical intervention programmed that could interfere with the physical exercise program.

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Frailty status or Physical Function change (composite outcome) | 8 months
  Frailty will be determined with the Frailty Phenotype and Physical Function with the SPPB

SECONDARY OUTCOMES:
Hospitalization | 1 year
  Number of hospitalizations during the follow-up for any cause.
Emergency department visits | 1 year
  Number of visits during the follow-up for any cause.
Mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on request. Study protocol, statistical analysis and clinical study report will be shared when data will be published in a Journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: At data Journal publication

REFERENCES:
- [Background] Kojima G, Iliffe S, Walters K. Frailty index as a predictor of mortality: a systematic review and meta-analysis. Age Ageing. 2018 Mar 1;47(2):193-200. doi: 10.1093/ageing/afx162. PMID 29040347
- [Background] Hoogendijk EO, Romero L, Sanchez-Jurado PM, Flores Ruano T, Vina J, Rodriguez-Manas L, Abizanda P. A New Functional Classification Based on Frailty and Disability Stratifies the Risk for Mortality Among Older Adults: The FRADEA Study. J Am Med Dir Assoc. 2019 Sep;20(9):1105-1110. doi: 10.1016/j.jamda.2019.01.129. Epub 2019 Mar 8. PMID 30853426
- [Background] Abizanda P, Romero L, Sanchez-Jurado PM, Martinez-Reig M, Gomez-Arnedo L, Alfonso SA. Frailty and mortality, disability and mobility loss in a Spanish cohort of older adults: the FRADEA study. Maturitas. 2013 Jan;74(1):54-60. doi: 10.1016/j.maturitas.2012.09.018. Epub 2012 Oct 26. PMID 23107816
- [Background] Kojima G. Frailty as a Predictor of Nursing Home Placement Among Community-Dwelling Older Adults: A Systematic Review and Meta-analysis. J Geriatr Phys Ther. 2018 Jan/Mar;41(1):42-48. doi: 10.1519/JPT.0000000000000097. PMID 27341327
- [Background] Kojima G. Frailty as a predictor of hospitalisation among community-dwelling older people: a systematic review and meta-analysis. J Epidemiol Community Health. 2016 Jul;70(7):722-9. doi: 10.1136/jech-2015-206978. Epub 2016 Mar 1. PMID 26933121
- [Background] Apostolo J, Cooke R, Bobrowicz-Campos E, Santana S, Marcucci M, Cano A, Vollenbroek-Hutten M, Germini F, D'Avanzo B, Gwyther H, Holland C. Effectiveness of interventions to prevent pre-frailty and frailty progression in older adults: a systematic review. JBI Database System Rev Implement Rep. 2018 Jan;16(1):140-232. doi: 10.11124/JBISRIR-2017-003382. PMID 29324562
- [Background] Tarazona-Santabalbina FJ, Gomez-Cabrera MC, Perez-Ros P, Martinez-Arnau FM, Cabo H, Tsaparas K, Salvador-Pascual A, Rodriguez-Manas L, Vina J. A Multicomponent Exercise Intervention that Reverses Frailty and Improves Cognition, Emotion, and Social Networking in the Community-Dwelling Frail Elderly: A Randomized Clinical Trial. J Am Med Dir Assoc. 2016 May 1;17(5):426-33. doi: 10.1016/j.jamda.2016.01.019. Epub 2016 Mar 3. PMID 26947059
- [Derived] Abizanda Saro A, Garcia Molina R, Alcantud Corcoles R, Maestre Moreno M, Sanchez Uceda R, Moron Merchante I, Aragones Jimenez A, Gonzalez Cespedes MD, Montero Alia P, Simarro Rueda M, Torres Anton L, Martinez Garcia P, Soriano Fernandez H, Corcoles Garcia M, Reyes Abreu AM, Morcillo Gonzalez MN, Garcia Paez E, Rodriguez Sanchez B, Saez Blesa M, Cortes Zamora EB, Andres Pretel F, Avendano Cespedes A; FRAILMERIT Study Group; Abizanda P. Efficacy of a Multicomponent Intervention for Frailty or Physical Function in Prefrail or Frail Older Adults: FRAILMERIT Multicenter Clinical Trial. J Am Geriatr Soc. 2025 Dec 28. doi: 10.1111/jgs.70266. Online ahead of print. PMID 41456342